CLINICAL TRIAL: NCT04186806
Title: An Evaluation of the Efficacy of 3M Dry Mouth Moisturizing Spray on the Relief of Dry Mouth Symptoms
Brief Title: Evaluation of the Efficacy of 3M Dry Mouth Moisturizing Spray
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EM-11-050038
Record Dates: First submitted 2019-10-08; First posted 2019-12-05 (Actual); Results first posted 2020-11-20 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Intervention Model Description: All subjects completing the wash-in procedures and meeting inclusion/exclusion criteria will undergo a pre-study 5-hour visit (the day before randomization) to assess the effect of water on their dry mouth symptoms. The subjects will return the next day for confirmation that inclusion/exclusion criteria and the wash-in procedures continue to be met or followed. Eligible subjects will be randomized at this baseline visit in a 1:1 ratio to one of two treatment orders: A->B (AB) or B->A (BA).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- 3M Dry Mouth Moisturizing Spray (Experimental): Dry mouth agent
  Interventions: Device: 3M Dry Mouth Moisturizing Spray to Biotene Moisturizing Mouth Spray; Device: Biotene Moisturizing Mouth Spray to 3M Dry Mouth Moisturizing Spray
- Biotene Moisturizing Mouth Spray (Active Comparator): Dry mouth agent
  Interventions: Device: 3M Dry Mouth Moisturizing Spray to Biotene Moisturizing Mouth Spray; Device: Biotene Moisturizing Mouth Spray to 3M Dry Mouth Moisturizing Spray

INTERVENTIONS:
Device: 3M Dry Mouth Moisturizing Spray to Biotene Moisturizing Mouth Spray — 20 ml bottle
Device: Biotene Moisturizing Mouth Spray to 3M Dry Mouth Moisturizing Spray — 44.3 ml bottle

SUMMARY:
The purpose of the clinical trial is to evaluate and validate the performance of the experimental mouth spray when used by persons with mild to severe dry mouth symptoms.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the efficacy of 3M Dry Mouth Moisturizing Spray to reduce symptoms of dry mouth for up to 4 hours and after 7 days of use. In addition, this study aims to support comparative claims.

ELIGIBILITY:
Inclusion Criteria:

Screening - Start of Wash-In Visit

* Subject who is ≥18 years of age and complains of dry mouth
* Only 1 subject per household is allowed into study
* Subject with a Challacombe scale score of 1 or higher
* Subject agrees to refrain from eating spicy foods and foods containing garlic beginning 48-hours prior to all study visits
* Subject agrees to eat a meal prior to all study visits that include sample evaluation in the clinic
* Subject agrees to not eat, drink, chew tobacco, chew gum, smoke, brush or floss teeth for 2-hours prior to sample evaluation study visits
* Subject agree to not use any oral care products and any type of breath mint or lozenges for 2-hours prior to sample evaluation study visits
* Subject agrees to refrain from any food and liquid during the 5-hour study visits except for what is provided by the study research staff (e.g., water and treatments A and B during evaluation periods)
* Subject agrees to only use those clinical oral care supplies provided during the entire study
* Able to understand and willing to sign the Informed Consent Form

Water Only Evaluation Visit

* Subject has successfully completed a ≥ 2-day wash-in period
* Subject has Challacombe scale score of 1 or higher
* Subject has refrained from eating spicy foods and foods containing garlic beginning 48-hours prior to the sample evaluation visits
* Subject ate a meal prior to sample evaluation study visits
* Subject has not eaten, drank, chewed tobacco, chewed gum, smoked, brushed or flossed teeth for 2-hours prior to sample evaluation study visits
* Subject has not used any oral care products, any type of breath mint or lozenges for 2-hours prior to sample evaluation study visits
* Subject agrees to refrain from any food and liquid during the 5-hour study visits except for what is provided by the study research staff (e.g., water and treatments A and B during evaluation periods)
* Subject has used only those clinical oral care supplies provided during study

Baseline Period 1/Randomization Visit

* Subject has successfully completed a ≥ 2-day wash-in period
* Subject has a Challacombe Scale score of 1 or higher
* Subject has refrained from eating spicy foods and foods containing garlic beginning 48-hours prior to sample evaluation study visits
* Subject ate a meal prior to sample evaluation study visits
* Subject has not eaten, drank, chewed tobacco, chewed gum, smoked, brushed or flossed teeth for 2-hours prior to sample evaluation study visits
* Subject has not used any oral care products and any type of breath mint or lozenges for 2-hours prior to sample evaluation study visits
* Subject agrees to refrain from any food and liquid during the 5-hour study visits except for what is provided by the study research staff (e.g., water and treatments A and B during evaluation periods)
* Subject has used only those clinical oral care supplies provided during study

Exclusion Criteria:

Subject Exclusion Criteria for Start of Wash-In, Water Only Evaluation and Baseline Period 1 (Randomization Visit)

* Subject has active mouth sores (e.g., cold sores, cuts, burns, canker sores)
* Subject has a life-threatening pathological condition
* Subject is participating in another clinical trial at the time of the study
* Subject has profound marginal periodontal disease (purulent exudate, tooth mobility, and/or extensive alveolar bone loss)
* Medical and oral conditions that, in the investigator's judgment, may compromise the subject's safety or interfere with the conduct and outcome of the study
* Difficult to be compliant with recalls, such as extensive travel commitments, lack of transportation etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-02 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Li, DDS,MSD,PhD, Principal Investigator — Loma Linda University, School of Dentistry
Locations (1):
- Loma Linda University, School of Dentistry, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Locker D. Xerostomia in older adults: a longitudinal study. Gerodontology. 1995 Jul;12(1):18-25. doi: 10.1111/j.1741-2358.1995.tb00125.x. PMID 8626175
- [Background] Fox PC. Management of dry mouth. Dent Clin North Am. 1997 Oct;41(4):863-75. PMID 9344281
- [Background] Guijarro Guijarro B, Lopez Sanchez AF, Hernandez Vallejo G. Treatment of xerostomia. A review. Med Oral. 2001 Jan-Feb;6(1):7-18. English, Spanish. PMID 11488135
- [Background] Fontana M, Zunt S, Eckert GJ, Zero D. A screening test for unstimulated salivary flow measurement. Oper Dent. 2005 Jan-Feb;30(1):3-8. PMID 15765951
- [Background] Andersson G, Johansson G, Attstrom R, Edwardsson S, Glantz PO, Larsson K. Comparison of the effect of the linseed extract Salinum and a methyl cellulose preparation on the symptoms of dry mouth. Gerodontology. 1995 Jul;12(1):12-7. doi: 10.1111/j.1741-2358.1995.tb00124.x. PMID 8626174

RESULTS

PARTICIPANT FLOW:
Groups:
- 3M Dry Mouth Moisturizing Spray Then Biotene Moisturizing Mouth Spray: Dry Mouth Agent: 3M Dry Mouth Moisturizing Spray: 20 ml bottle
  or
  Dry Mouth Agent: Biotene Moisturizing Mouth Spray: 44 ml bottle
- Biotene Moisturizing Mouth Spray Then 3M Dry Mouth Moisturizing Spray: Dry mouth agent: Biotene Moisturizing Mouth Spray: 44 ml bottle
  or
  Dry mouth agent: 3M Dry Mouth Moisturizing Spray: 20 ml bottle
Period: Period 1: 7 Days
Arm/Group | 3M Dry Mouth Moisturizing Spray Then Biotene Moisturizing Mouth Spray | Biotene Moisturizing Mouth Spray Then 3M Dry Mouth Moisturizing Spray
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout Period: at Least 2 Days
Arm/Group | 3M Dry Mouth Moisturizing Spray Then Biotene Moisturizing Mouth Spray | Biotene Moisturizing Mouth Spray Then 3M Dry Mouth Moisturizing Spray
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0
Period: Period 2: 7 Days
Arm/Group | 3M Dry Mouth Moisturizing Spray Then Biotene Moisturizing Mouth Spray | Biotene Moisturizing Mouth Spray Then 3M Dry Mouth Moisturizing Spray
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 3M Spray Then Biotene Spray: 3M Dry Mouth Moisturizing Spray then Biotene Dry Mouth Moisturizing Spray
- Biotene Spray Then 3M Spray: Biotene Dry Mouth Moisturizing Spray then 3M Dry Mouth Moisturizing Spray
- Total: Total of all reporting groups
Arm/Group | 3M Spray Then Biotene Spray | Biotene Spray Then 3M Spray | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (13.67) | 49.7 (14.88) | 49.4 (14.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 11 | 18
  Not Hispanic or Latino | 13 | 9 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 2 | 3
  White | 16 | 15 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40
Currently using Dry Mouth Products [Count of Participants; unit: Participants]
  Currently using dry mouth products | 2 | 2 | 4
  Not currently using dry mouth products | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: 10 cm Mouth Dryness Visual Analog Score
Description: Primary endpoint will be paired-difference in Visual Analog Scale (VAS) between experimental and active control product. On the scale 0 represents normal and 10 represents worst imaginable dry mouth symptoms.
Time Frame: 15 minutes post dose
Population: Intent to treat (ITT) with Group Means Imputation
Measure: Mean (Standard Deviation); unit: cm
Groups:
- 3M(TM) Dry Mouth Moisturizing Spray: Dry mouth agent
  3M(TM) Dry Mouth Moisturizing Spray: 20 ml bottle
  Distilled water: 15 ml
- Biotene Moisturizing Mouth Spray: Dry mouth agent
  Biotene Moisturizing Mouth Spray: 44.3 ml bottle
  Distilled water: 15 ml
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 40
cm | 4.51 (2.228) | 4.6 (2.604)
Statistical Analysis 1: Comparison: 3M(TM) Dry Mouth Moisturizing Spray vs Biotene Moisturizing Mouth Spray; Test type: Non-Inferiority — Non-inferiority margin was 1.5 cm; Mixed Models Analysis — The conclusion of the non-inferiority test is based on the 95% confidence interval and not on a p value. A p value was not computed; Mean Difference (Final Values) = -0.3426, 95% CI 2-sided [-1.2601 to 0.5749] — Non-inferiority testing was carried out using 95% confidence intervals

2. Secondary Outcome: 10 cm Mean Mouth Dryness Visual Analog Score
Description: Mean Visual Analog Scale (VAS) on the scale 0 represents normal and 10 represents worst imaginable dry mouth symptoms
Time Frame: 240 minutes post dose
Population: Intent to Treat (ITT) with Group Means Imputation
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 40
cm | 5.14 (1.689) | 5.68 (2.261)

3. Secondary Outcome: 10 cm Mouth Dryness Visual Analog Score
Description: Paired-difference Visual Analog Scale (VAS) between both experimental and active control against water control. The range of possible values is -10 to +10. A negative value means is a better outcome than water. A positive value means is a worse outcome than water.
Time Frame: 240 minutes
Population: Intent to Treat (ITT) with Group Means Imputation
Measure: Least Squares Mean (Standard Error); unit: cm
Groups:
- 3M Dry Mouth Moisturizing Spray: Dry mouth agent
  3M Dry Mouth Moisturizing Spray: 20 ml bottle
  Distilled water: 15 ml
Arm/Group | 3M Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 40
cm | -2.322 (0.3115) | -1.665 (0.3576)

4. Secondary Outcome: 10 cm Mean Mouth Dryness Visual Analog Score
Description: Mean Visual Analog Scale (VAS) on the scale 0 represents normal and 10 represents worst imaginable dry mouth symptoms
Time Frame: 5 minutes
Population: Intent to Treat (ITT) with Group Means Imputation
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 40
cm | 4.54 (2.128) | 4.62 (2.703)

5. Secondary Outcome: 10 cm Mean Mouth Dryness Visual Analog Scale
Description: Mean Visual Analog Scale (VAS) on the scale 0 represents normal and 10 represents worst imaginable dry mouth symptoms
Time Frame: 30 minutes
Population: Intent to Treat (ITT) with Group Means Imputation
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 40
cm | 4.51 (2.172) | 4.75 (2.403)

6. Secondary Outcome: 10 cm Mean Mouth Dryness Visual Analog Scale
Description: Mean Visual Analog Scale (VAS) on the scale 0 represents normal and 10 represents worst imaginable dry mouth symptoms
Time Frame: 60 minutes
Population: Intent to Treat (ITT) with Group Means Imputation
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 40
cm | 4.58 (2.092) | 5.04 (2.168)

7. Secondary Outcome: 10 cm Mean Mouth Dryness Visual Analog Scale
Description: Mean Visual Analog Scale (VAS) on the scale 0 represents normal and 10 represents worst imaginable dry mouth symptoms
Time Frame: 120 minutes
Population: Intent to Treat (ITT) with Group Means Imputation
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 40
cm | 4.86 (1.832) | 5.41 (2.143)

8. Secondary Outcome: 10 cm Mouth Dryness Visual Analog Scale
Description: as for outcome 3
Time Frame: 5 minutes
Population: Intent to Treat (ITT) with Group Means Imputation
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 40
cm | -2.203 (0.3042) | -1.871 (0.3780)

9. Secondary Outcome: 10 cm Mouth Dryness Visual Analog Scale
Description: as for outcome 3
Time Frame: 15 minutes
Population: Intent to Treat (ITT) with Group Means Imputation
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 40
cm | -2.394 (0.3095) | -2.036 (0.3476)

10. Secondary Outcome: 10 cm Mouth Dryness Visual Analog Scale
Description: as for outcome 3
Time Frame: 30 minutes
Population: Intent to Treat (ITT) with Group Means Imputation
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 40
cm | -2.420 (0.3111) | -1.900 (0.3176)

11. Secondary Outcome: 10 cm Mouth Dryness Visual Analog Score
Description: as for outcome 3
Time Frame: 60 minutes
Population: Intent to Treat (ITT) with Group Means Imputation
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 40
cm | -2.455 (0.3172) | -1.833 (0.3090)

12. Secondary Outcome: 10 cm Mouth Dryness Visual Analog Score
Description: as for outcome 3
Time Frame: 120 minutes
Population: Intent to Treat (ITT) with Group Means Imputation
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 40
cm | -2.364 (0.3108) | -1.657 (0.3281)

13. Secondary Outcome: Response on Dry Mouth Relief
Description: Count of each category of the ordinal scale 0 = No Relief and 4 = Significant/Excellent
Time Frame: 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  0=No Relief | 3 | 3
  1=Not Enough | 4 | 6
  2=Some/Good | 14 | 16
  3=Very Good | 13 | 6
  4=Significant/Excellent | 6 | 8

14. Secondary Outcome: Response on Dry Mouth Relief
Description: Count of each category of the ordinal scale 0 = No Relief and 4 = Significant/Excellent
Time Frame: 15 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  0=No Relief | 2 | 3
  1=Not Enough | 7 | 4
  2=Some/Good | 10 | 19
  3=Very Good | 16 | 8
  4=Significant/Excellent | 5 | 5

15. Secondary Outcome: Response on Dry Mouth Relief
Description: Count of each category of the ordinal scale 0 = No Relief and 4 = Significant/Excellent
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  0=No Relief | 2 | 3
  1=Not Enough | 6 | 6
  2=Some/Good | 13 | 21
  3=Very Good | 17 | 8
  4=Significant/Excellent | 2 | 1

16. Secondary Outcome: Response on Dry Mouth Relief
Description: Count of each category of the ordinal scale 0 = No Relief and 4 = Significant/Excellent
Time Frame: 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  0=No Relief | 3 | 4
  1=Not Enough | 5 | 5
  2=Some/Good | 18 | 22
  3=Very Good | 13 | 7
  4=Significant/Excellent | 1 | 1

17. Secondary Outcome: Response on Dry Mouth Relief
Description: Count of each category of the ordinal scale 0 = No Relief and 4 = Significant/Excellent
Time Frame: 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  0=No Relief | 3 | 4
  1=Not Enough | 10 | 14
  2=Some/Good | 15 | 15
  3=Very Good | 11 | 5
  4=Significant/Excellent | 1 | 1

18. Secondary Outcome: Response on Dry Mouth Relief
Description: Count of each category of the ordinal scale 0 = No Relief and 4 = Significant/Excellent
Time Frame: 240 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  0=No Relief | 6 | 6
  1=Not Enough | 13 | 16
  2=Some/Good | 12 | 11
  3=Very Good | 9 | 5
  4=Significant/Excellent | 0 | 1

19. Secondary Outcome: Response to Effectively Lubricates the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 2 | 3
  2= Fair | 7 | 8
  3= Good | 10 | 16
  4= Very Good | 14 | 4
  5= Excellent | 7 | 8

20. Secondary Outcome: Response to Effectively Lubricates the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 15 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 2 | 3
  2= Fair | 8 | 7
  3= Good | 10 | 17
  4= Very Good | 15 | 6
  5= Excellent | 5 | 6

21. Secondary Outcome: Response to Effectively Lubricates the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 2 | 3
  2= Fair | 9 | 12
  3= Good | 13 | 15
  4= Very Good | 15 | 8
  5= Excellent | 1 | 1

22. Secondary Outcome: Response to Effectively Lubricates the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 4 | 3
  2= Fair | 11 | 15
  3= Good | 14 | 13
  4= Very Good | 10 | 7
  5= Excellent | 1 | 1

23. Secondary Outcome: Response to Effectively Lubricates the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 5 | 9
  2= Fair | 15 | 12
  3= Good | 12 | 12
  4= Very Good | 7 | 5
  5= Excellent | 1 | 1

24. Secondary Outcome: Response to Effectively Lubricates the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 240 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 9 | 9
  2= Fair | 14 | 18
  3= Good | 10 | 6
  4= Very Good | 6 | 4
  5= Excellent | 1 | 2

25. Secondary Outcome: Response to Feel Comfortable in the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 1 | 2
  2= Fair | 5 | 7
  3= Good | 13 | 15
  4= Very Good | 11 | 6
  5= Excellent | 10 | 9

26. Secondary Outcome: Response to Feel Comfortable in the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 15 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 1 | 2
  2= Fair | 5 | 6
  3= Good | 14 | 16
  4= Very Good | 13 | 8
  5= Excellent | 7 | 7

27. Secondary Outcome: Response to Feel Comfortable in the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 1 | 3
  2= Fair | 6 | 6
  3= Good | 14 | 20
  4= Very Good | 16 | 6
  5= Excellent | 3 | 4

28. Secondary Outcome: Response to Feel Comfortable in the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 2 | 3
  2= Fair | 9 | 11
  3= Good | 15 | 13
  4= Very Good | 11 | 10
  5= Excellent | 3 | 2

29. Secondary Outcome: Response to Feel Comfortable in the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 4 | 4
  2= Fair | 14 | 11
  3= Good | 10 | 14
  4= Very Good | 9 | 8
  5= Excellent | 3 | 2

30. Secondary Outcome: Response to Feel Comfortable in the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 240 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 5 | 6
  2= Fair | 14 | 14
  3= Good | 12 | 11
  4= Very Good | 6 | 5
  5= Excellent | 3 | 3

31. Secondary Outcome: Response to Soothing in the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 1 | 1
  2= Fair | 6 | 7
  3= Good | 10 | 16
  4= Very Good | 12 | 6
  5= Excellent | 11 | 9

32. Secondary Outcome: Response to Soothing in the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 15 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 1 | 1
  2= Fair | 7 | 8
  3= Good | 11 | 17
  4= Very Good | 13 | 6
  5= Excellent | 8 | 7

33. Secondary Outcome: Response to Soothing in the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 1 | 2
  2= Fair | 8 | 12
  3= Good | 14 | 15
  4= Very Good | 13 | 8
  5= Excellent | 4 | 2

34. Secondary Outcome: Response to Soothing in the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 3 | 3
  2= Fair | 10 | 12
  3= Good | 13 | 15
  4= Very Good | 12 | 7
  5= Excellent | 2 | 2

35. Secondary Outcome: Response to Soothing in the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 4 | 7
  2= Fair | 14 | 11
  3= Good | 12 | 13
  4= Very Good | 8 | 6
  5= Excellent | 2 | 2

36. Secondary Outcome: Response to Soothing in the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 240 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 7 | 8
  2= Fair | 16 | 15
  3= Good | 8 | 9
  4= Very Good | 7 | 4
  5= Excellent | 2 | 3

37. Secondary Outcome: Response to Effectively Moistens the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 3 | 3
  2= Fair | 5 | 6
  3= Good | 11 | 17
  4= Very Good | 12 | 5
  5= Excellent | 9 | 8

38. Secondary Outcome: Response to Effectively Moistens the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 15 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 2 | 3
  2= Fair | 7 | 6
  3= Good | 12 | 18
  4= Very Good | 12 | 6
  5= Excellent | 7 | 6

39. Secondary Outcome: Response to Effectively Moistens the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 3 | 3
  2= Fair | 7 | 9
  3= Good | 14 | 19
  4= Very Good | 13 | 7
  5= Excellent | 3 | 1

40. Secondary Outcome: Response to Effectively Moistens the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 5 | 3
  2= Fair | 11 | 12
  3= Good | 13 | 15
  4= Very Good | 9 | 8
  5= Excellent | 2 | 1

41. Secondary Outcome: Response to Effectively Moistens the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 6 | 8
  2= Fair | 16 | 15
  3= Good | 9 | 9
  4= Very Good | 8 | 6
  5= Excellent | 1 | 1

42. Secondary Outcome: Response to Effectively Moistens the Mouth
Description: 5 point ordinal scale 1 = Poor and 5 = Excellent
Time Frame: 240 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
Number analyzed (Participants) | 40 | 39
Participants
  1= Poor | 12 | 8
  2= Fair | 12 | 20
  3= Good | 8 | 5
  4= Very Good | 8 | 4
  5= Excellent | 0 | 2

ADVERSE EVENTS:
Time Frame: For the entire 7 day treatment period for each study arm
Arm/Group | 3M(TM) Dry Mouth Moisturizing Spray | Biotene Moisturizing Mouth Spray
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/39
Other Adverse Events (participants affected / at risk) | 7/40 | 7/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3M(TM) Dry Mouth Moisturizing Spray (N=40) | Biotene Moisturizing Mouth Spray (N=39)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Abdominal Skin Sore
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3M(TM) Dry Mouth Moisturizing Spray (N=40) | Biotene Moisturizing Mouth Spray (N=39)
Aphthous Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hypoesthesia Oral (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral Discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oropharyngeal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paresthesia Oral (Gastrointestinal disorders) | 1 (1) | 2 (2)
Salivary Hypersecretion (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT04186806/Prot_SAP_000.pdf